CLINICAL TRIAL: NCT00141492
Title: A Double Blind, Randomized, Placebo-Controlled, Parallel Study to Evaluate the Efficacy and Safety of Androgel, as an Adjunct to Hypoglycemic Therapy, in the Treatment of Hypogonadal and Low Testosterone Men With Type 2 Diabetes
Brief Title: Efficacy and Safety of Androgel in the Treatment of Hypogonadal and Low Testosterone Men With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S176.2.101
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Type 2 Diabetes; Hypogonadism
Keywords: Type 2 diabetes; hypogonadism; testosterone; glycosylated hemoglobin A1C
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypogonadism | interventions — Testosterone

INTERVENTIONS:
Drug: Androgel (testosterone gel)

SUMMARY:
This study is to investigate how well Androgel, when tested against placebo gel, helps to control blood sugar levels in males with type 2 diabetes who have low testosterone (the main male hormone) blood levels and are taking oral diabetic medicines alone or in combination with insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and write
2. Males
3. Between 30-80 years old
4. Have type 2 diabetes
5. Diagnoses of hypogonadism or low testosterone

Exclusion Criteria:

1. On insulin monotherapy
2. Use of testosterone therapy within the last 6 months
3. Male breast cancer
4. History of prostate cancer
5. History of clinically significant sleep apnea

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (70):
- United States (70):
  - Site 58, Birmingham, Alabama
  - Site 67, Calera, Alabama
  - Site 54, Mobile, Alabama
  - Site 16, Phoenix, Arizona
  - Site 35, Anaheim, California
  - Site 23, Concord, California
  - Site 55, La Jolla, California
  - Site 8, Los Gatos, California
  - Site 12, Mission Viejo, California
  - Site 1, Torrance, California
  - Site 25, Glastonbury, Connecticut
  - Site 13, Fort Lauderdale, Florida
  - Site 43, Jacksonville, Florida
  - Site 33, Ocala, Florida
  - Site 27, Tampa, Florida
  - Site 21, West Palm Beach, Florida
  - Site 7, Atlanta, Georgia
  - Site 26, Columbus, Georgia
  - Site 29, Boise, Idaho
  - Site 45, Idaho Falls, Idaho
  - Site 51, Chicago, Illinois
  - Site 32, Des Moines, Iowa
  - Site 5, Baton Rouge, Louisiana
  - Site 70, Baltimore, Maryland
  - Site 9, Springfield, Massachusetts
  - Site 48, Watertown, Massachusetts
  - Site 19, Detroit, Michigan
  - Site 61, Livonia, Michigan
  - Site 40, Tupelo, Mississippi
  - Site 65, Chesterfield, Missouri
  - Site 15, Kansas City, Missouri
  - Site 41, Omaha, Nebraska
  - Site 34, Las Vegas, Nevada
  - Site 24, Jersey City, New Jersey
  - Site 49, Buffalo, New York
  - Site 71, New York, New York
  - Site 44, Fayetteville, North Carolina
  - Site 28, Morehead City, North Carolina
  - Site 60, Morehead City, North Carolina
  - Site 31, Portland, Oregon
  - Site 3, Portland, Oregon
  - Site 68, Altoona, Pennsylvania
  - Site 4, Bala-Cynwyd, Pennsylvania
  - Site 64, Carlisle, Pennsylvania
  - Site 38, Lansdale, Pennsylvania
  - Site 46, Shippensburg, Pennsylvania
  - Site 14, Greer, South Carolina
  - Site 20, Arlington, Texas
  - Site 11, Dallas, Texas
  - Site 10, Houston, Texas
  - Site 18, Houston, Texas
  - Site 2, Houston, Texas
  - Site 36, Houston, Texas
  - Site 39, Houston, Texas
  - Site 42, Houston, Texas
  - Site 47, Houston, Texas
  - Site 53, Houston, Texas
  - Site 62, Houston, Texas
  - Site 63, Houston, Texas
  - Site 69, Houston, Texas
  - Site 6, Humble, Texas
  - Site 30, La Porte, Texas
  - Site 66, Midland, Texas
  - Site 37, San Antonio, Texas
  - Site 56, Sugarland, Texas
  - Site 57, Sugarland, Texas
  - Site 52, Ogden, Utah
  - Site 17, Salt Lake City, Utah
  - Site 22, Salem, Virginia
  - Site 50, Seattle, Washington